CLINICAL TRIAL: NCT02376530
Title: Price Changes and Nutrient Profiling Among Adult Grocery Shoppers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leonard Epstein, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 1101757-1-60725
Record Dates: First submitted 2014-07-18; First posted 2015-03-03 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Nutrition; Food Purchases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual shopping (No Intervention): No change in condition.
- Nutrient profiling (Experimental): Nutrient profiling system will be present during shopping session.
  Interventions: Behavioral: Nutrient profiling
- Price change (Experimental): Price changes will be present during shopping session.
  Interventions: Behavioral: Price Changes
- Nutrient profiling and price change (Experimental): Nutrient profiling system and price changes will be present during shopping session.
  Interventions: Behavioral: Nutrient profiling; Behavioral: Price Changes

INTERVENTIONS:
Behavioral: Nutrient profiling — Nutrient profiling system will be present during shopping session.
  Arms: Nutrient profiling; Nutrient profiling and price change
Behavioral: Price Changes — Price changes will be present during shopping session.
  Arms: Nutrient profiling and price change; Price change

SUMMARY:
The purpose of the research is to examine the association between price changes, nutrient profiling, and grocery food purchases among household grocery shoppers.

DETAILED DESCRIPTION:
Participants will be asked to select a week's worth of groceries for their household from a virtual online grocery store. Shoppers will be randomly assigned to one of four conditions (control, nutrient profiling, price change, nutrient profiling and price change).

ELIGIBILITY:
Inclusion Criteria:

* primary household grocery shopper
* at least 19 years old
* one or more child (2-18yrs) living full time in the household

Exclusion Criteria:

* not the primary household grocery shopper
* no dietary, medical, or psychopathology conditions that could interfere with the study
* under the age 19
* no children (2-18yrs) living full time in the household

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 788 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Epstein, Ph.D, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Division of Behavioral Medicine, University at Buffalo — http://medicine.buffalo.edu/departments/pediatrics/divisions/behavioral-medicine.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the WNY community between 2012-2014.
Period: Overall Study
Arm/Group | Usual Shopping | Nutrient Profiling | Price Change | Nutrient Profiling and Price Change
Started | 196 | 198 | 197 | 197
Completed | 196 | 198 | 197 | 197
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Shopping | Nutrient Profiling | Price Change | Nutrient Profiling and Price Change | Total
Number analyzed (Participants) | 196 | 198 | 197 | 197 | 788
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (8.6) | 42.5 (8.8) | 42.4 (8.2) | 41.6 (7.8) | 42.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 198 | 197 | 197 | 788
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 12 | 8 | 11 | 38
  Not Hispanic or Latino | 188 | 185 | 188 | 185 | 746
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 2 | 5
  Asian | 2 | 5 | 2 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 2
  Black or African American | 44 | 39 | 47 | 39 | 169
  White | 135 | 140 | 140 | 140 | 555
  More than one race | 9 | 8 | 3 | 5 | 25
  Unknown or Not Reported | 5 | 4 | 4 | 7 | 20
Region of Enrollment [Number; unit: participants]
  United States | 196 | 198 | 197 | 197 | 788
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 31.0 (8.0) | 30.8 (7.9) | 30.9 (8.2) | 31.3 (8.7) | 31.0 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Nutritional Quality of Food Purchases
Description: The Overall Nutrient Quality Index (ONQI) was used to assess nutritional quality of foods purchased. The ONQI is a 1 - 100 scale in which higher numbers indicate higher nutritional quality. Each food is given a score based on a ratio with positive health nutrients in the numerator and detrimental health nutrients in the denominator, based on a proprietary algorithm created by NuVal. The average ONQI score for all the groceries purchases was used as the outcome measure, of ONQI scores on a scale.
Time Frame: Participants were followed for one shopping session, an average of 2.5 hours
Population: Data was analyzed for 781 participants. Two participants did not understand the study, 2 participants had incorrect price manipulations during their session, 1 participant was ill during the session, 1 participant had her young daughter in the room during the experiment and 1 participant did not have a household to shop for.
Measure: Least Squares Mean (Standard Deviation); unit: Average NUVAL Score
Arm/Group | Usual Shopping | Nutrient Profiling | Price Change | Nutrient Profiling and Price Change
Number analyzed (Participants) | 193 | 197 | 196 | 195
Average NUVAL Score | 37.62 (14.84) | 41.12 (15.06) | 39.66 (13.30) | 41.01 (14.21)

ADVERSE EVENTS:
Arm/Group | Usual Shopping | Nutrient Profiling | Price Change | Nutrient Profiling and Price Change
Serious Adverse Events (participants affected / at risk) | 0/196 | 0/198 | 0/197 | 0/197
Other Adverse Events (participants affected / at risk) | 0/196 | 0/198 | 0/197 | 0/197

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No